CLINICAL TRIAL: NCT03972137
Title: Development and Pilot Investigation of Heart Rate Variability Biofeedback for Smoking Cessation
Brief Title: Heart Rate Variability Biofeedback for Smoking Cessation
Acronym: HRVB-SCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Teresa M. Leyro, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018001848; R34DA043751 (NIH)
Record Dates: First submitted 2019-05-20; First posted 2019-06-03 (Actual); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Tobacco Smoking
Keywords: Smoking Cessation; Heart rate variability biofeedback
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation | interventions — Cognitive Behavioral Therapy; Biofeedback, Psychology; Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: All participants received individualized smoking cessation therapy (SCT), nicotine replacement therapy patch (NRT) and heart rate variability biofeedback (HRVB).
Masking Description: This is an open trial with all participants receiving what will become the 'active intervention' in a subsequent randomized clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Heart Rate Variability Biofeedback-Smoking Cessation Therapy (Experimental): All participants in this open trial received individualized cognitive-behavioral smoking cessation treatment (SCT), up to 8 weeks of the transdermal nicotine patch (NRT) and individualized heart rate variability biofeedback (HRVB).
  Interventions: Behavioral: Cognitive-Behavioral Smoking Cessation; Behavioral: Heart Rate Variability Biofeedback (HRVB); Drug: Transdermal Nicotine patch

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Smoking Cessation — Participants were provided with six individualized smoking cessation counseling sessions designed to help them prepare to quit, set a quit date, behaviorally manage early abstinence, and to resume cessation upon lapse.
  Other Names: Cognitive-behavioral therapy; Smoking cessation counseling (SCT)
Behavioral: Heart Rate Variability Biofeedback (HRVB) — All participants were provided with individualized training in resonance breathing using biofeedback to help improve self-regulation.
  Other Names: Biofeedback; Respiratory biofeedback
Drug: Transdermal Nicotine patch — All participants were offered up to eight weeks of transdermal nicotine patch, beginning on their quit date.
  Other Names: Nicotine patch; Nicotine replacement therapy (NRT)

SUMMARY:
Open trial of heart rate variability biofeedback as an adjunct to individualized smoking cessation counseling (SCT) plus transdermal nicotine replacement patch (NRT) in smokers with elevated emotional distress.

DETAILED DESCRIPTION:
The investigators propose to develop and pilot test heart rate variability biofeedback (HRVB) for smokers with elevated emotional distress as an adjunct to individual smoking cessation counseling (SCT) and transdermal nicotine patch (NRT). In this open trial, all participants received the active intervention. Findings will be used to refine the protocol in advance of a subsequent Phase III randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Smoking ≥5 cigarettes, daily, for at least two years
* expired carbon monoxide analysis of breath sample ≥8 ppm
* elevated affective distress
* motivation to quit
* computer proficient

Exclusion Criteria:

* current use of other tobacco or nicotine products for recreation or to aid in cessation, use of pharmacological intervention for cessation, or current enrollment in a psychosocial intervention for smoking cessation
* endorsement of current or past psychotic or manic symptoms indicative of bipolar spectrum or schizophrenia spectrum disorders and/or current suicidal or homicidal ideation
* inability to provide written informed consent
* current evidence of another substance use disorder
* severe visual or hearing impairments
* self-reported medical condition or medication use that may be contraindicated for participation in a HRVB or confound autonomic parameters:
* self-reported medical issues of potential concern to nicotine patch users

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Leyro, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers, School of Arts and Sciences, One Spring Street, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
We currently have no plans to share individual participant data from this small open trial as it will be used to guide refinement of a subsequent larger randomized controlled trial.

REFERENCES:
- [Background] Leyro TM, Buckman JF, Bates ME. Theoretical implications and clinical support for heart rate variability biofeedback for substance use disorders. Curr Opin Psychol. 2019 Dec;30:92-97. doi: 10.1016/j.copsyc.2019.03.008. Epub 2019 Apr 2. PMID 31055246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the New Brunswick, New Jersey area via flyer postings, clinic referrals, and social media advertisements. The first participant was enrolled April 24, 2019 and the last participant was enrolled November 12, 2019.
Pre-assignment Details: The intervention occurred across 10 sessions. All participants received individualized heart rate variability biofeedback at each session, smoking cessation therapy during 6 of the sessions and 8 weeks of transdermal nicotine patches. Two of the twelve consented participants who attended the baseline visit were not eligible and were not enrolled.
Groups:
- Heart Rate Variability Biofeedback- Smoking Cessation Therapy: All participants in this open trial received individualized cognitive-behavioral smoking cessation treatment, up to 8 weeks of the transdermal nicotine patch, and individualized heart rate variability biofeedback.
  Cognitive-Behavioral Smoking Cessation: Participants were provided with six individualized smoking cessation counseling sessions designed to help them prepare to quit, set a quit date, behaviorally manage early abstinence, and to resume cessation upon lapse.
  Heart Rate Variability Biofeedback: All participants were provided with individualized training in resonance breathing using biofeedback to help improve self-regulation.
  Nicotine patch: All participants were offered up to eight weeks of transdermal nicotine patch, beginning on their quit date.
Period: Overall Study
Arm/Group | Heart Rate Variability Biofeedback- Smoking Cessation Therapy
Started | 10
Enrolled | 10
Treatment Completed | 6
Follow-up Completed | 4
Completed | 4
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Enrolled: Participants who were eligible and completed the Baseline session
Arm/Group | Enrolled
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Participant Attendance
Description: Number of intervention sessions attended out of 10 possible sessions.
Time Frame: 7 weeks
Population: Data on both the Intent-to-treat (ITT) N=10 participants who completed the baseline session and were enrolled in the study and the n=7 who received more than one Heart Rate Variability Biofeedback Session (HRVB) and one Smoking Cessation Treatment (SCT) session (i.e. which occurred during their first intervention appointment) are reported.
Measure: Mean (Standard Deviation); unit: Sessions
Groups:
- Intent-to-treat (ITT): Participants who completed their baseline session and were enrolled in the study
- Remained in Treatment Beyond One Session: Excluding n=3 participants who withdrew following one intervention session.
Arm/Group | Intent-to-treat (ITT) | Remained in Treatment Beyond One Session
Number analyzed (Participants) | 10 | 7
Sessions | 6.30 (4.08) | 8.71 (1.49)

2. Primary Outcome: Intervention Feasibility: Participant Ratings of Effectiveness
Description: Effectiveness was assessed via self-report ratings on four items assessing the intervention in terms of helping them quit and manage emotional distress, rated on a 0=completely disagree to 4=completely agree Likert-type scale. Higher scores on this scale are indicative of greater perceived intervention efficacy. Mean scores obtained following the first intervention session and 3-month follow-up session are reported.
Time Frame: Week 1 (i.e., treatment initiation) and Week 16 (i.e., 3-month follow-up)
Population: Of the N=10 participants who were enrolled in the study, n=9 completed this measure following their baseline appointment; n=4 attended their 3-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- First Session: Participants who attended their first intervention session
- 3-month Follow-up (3MFU): Participants who attended their 3-month follow-up session
Arm/Group | First Session | 3-month Follow-up (3MFU)
Number analyzed (Participants) | 9 | 4
score on a scale | 3.03 (0.83) | 3.19 (0.52)

3. Primary Outcome: Intervention Feasibility: Participant Ratings of Appropriateness
Description: Appropriateness was assessed via self-report ratings on two items assessing the intervention in terms of comprehension and fit, rated on a 0=completely disagree to 4=completely agree Likert-type scale. Higher scores on this scale are indicative of greater perceived intervention appropriateness. Mean scores obtained following the first intervention session and 3-month follow-up session are reported.
Time Frame: Week 1 (i.e., treatment initiation) and Week 16 (i.e., 3-month follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | First Session | 3-month Follow-up (3MFU)
Number analyzed (Participants) | 9 | 4
score on a scale | 3.61 (0.69) | 2.87 (0.75)

4. Primary Outcome: Intervention Feasibility: Participant Ratings of Ease of the Intervention
Description: Ease of the Intervention was assessed via self-report ratings on three items assessing ease of use and fit into daily lifestyle, rated on a 0=completely disagree to 4=completely agree Likert-type scale. Higher scores on this scale are indicative of greater perceived ease of the intervention and fit into daily lifestyle. Mean scores obtained following the first intervention session and 3-month follow-up session are reported.
Time Frame: Week 1 (i.e., treatment initiation) and Week 16 (i.e., 3-month follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 3-month Follow-up (3MFU): Participants that attended their 3-month follow-up session
Arm/Group | First Session | 3-month Follow-up (3MFU)
Number analyzed (Participants) | 9 | 4
score on a scale | 2.4 (0.84) | 1.58 (0.32)

5. Primary Outcome: Intervention Acceptability: Participant Ratings of Satisfaction and Liking
Description: Satisfaction and liking were assessed via self-report ratings on five items assessing satisfaction with learning the intervention, liking the intervention, breathing techniques, nicotine replacement, and recommending the intervention to friends, rated on a 0=completely disagree to 4=completely agree Likert-type scale. Higher scores on this scale are indicative of greater intervention acceptability. Mean scores obtained following the first intervention session and 3-month follow-up session are reported.
Time Frame: Week 1 (i.e., treatment initiation) and Week 16 (i.e., 3-month follow-up)
Population: Of the N=10 participants who were enrolled in the study, n=9 completed this measure following their baseline appointment; n=3 attended their 3-month follow-up and provided complete data for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | First Session | 3-month Follow-up (3MFU)
Number analyzed (Participants) | 9 | 3
score on a scale | 3.24 (0.71) | 3.52 (0.31)

6. Secondary Outcome: Number of Participants With Self-Reported Abstinence, Cotinine Verified Abstinence, and Carbon Monoxide Analysis of Breathe Sample (CO < 8ppm)
Description: Quit status was assessed on Quit day via self-reported abstinence and carbon monoxide analysis of breath sample (CO <8 ppm). Given carbon monoxide analysis of breath may not be a valid indicator of cessation within the first 24 hours, we suggest interpretation of this outcome on Quit day with caution.
  Sustained smoking cessation was evaluated at study termination (i.e., 3-month follow-up) via self-reported abstinence, carbon monoxide analysis ( CO <8 ppm), and salivary cotinine (<10 ng/mL).
Time Frame: Week 3 (i.e., Quit Date) and Week 16 (i.e., 3-month follow-up)
Population: Of the N=9 who were eligible and initiated treatment, n=7 attended their quit date and n=4 attended their 3-month follow-up.
Measure: Number; unit: participants
Groups:
- Quit Date: Participants who attended their Quit day session
Arm/Group | Quit Date | 3-month Follow-up (3MFU)
Number analyzed (Participants) | 7 | 4
participants
  Self-Reported abstinence | 6 | 4
  Cotinine verified abstinence | NA — Salivary cotinine was only collected at 3-month follow-up | 4
  CO <8 parts per million (PPM) | 2 | 4

7. Secondary Outcome: Cigarettes Smoked Per Day
Description: Cigarettes Smoked Per Day (CPD) assessed via the well established Timeline Followback calendar interview were used to measure changes in smoking behavior from Week 0 (i.e., Baseline) through Week 3 (i.e., Quit date) and Week 16 (i.e., 3-month follow-up).
Time Frame: Week 0 (i.e., baseline), Week 3 (i.e., Quit Date) and Week 16 (i.e., 3-month follow-up)
Population: Of the N=10 participants who were eligible and attended the baseline session, n=7 attended their quit date and n=4 attended their 3-month follow-up session
Measure: Mean (Standard Deviation); unit: Cigarettes smoked per day (CPD)
Groups:
- Baseline (BL): Mean CPD at baseline was determined by averaging the total number of cigarettes smoked per day for 30 the days prior to the participant's baseline session. Data reflect participants who attended their baseline session.
- Quit Date: Mean CPD at Quit date was determined by averaging the total number of cigarettes smoked on their Quit-day session. Data reflect participants who attended their Quit-day session.
- 3-month Follow-up (3MFU): Mean CPD at 3-Month Follow-up was determined by averaging the total number of cigarettes smoked during the 7 days prior to their 3MFU session. Data reflect participants who attended their 3MFU session.
Arm/Group | Baseline (BL) | Quit Date | 3-month Follow-up (3MFU)
Number analyzed (Participants) | 10 | 7 | 4
Cigarettes smoked per day (CPD) | 11.56 (6.03) | 0.14 (0.38) | 0 (0)
Statistical Analysis 1: Comparison: Baseline (BL) vs Quit Date; Test type: Other — A paired-samples t-test was conducted to compare changes in cigarettes smoked per day from Baseline (BL) to Quit Day; p = .003, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 11.42, 95% CI 2-sided [5.79 to 17.05], Standard Deviation 6.08 — Mean difference represents the difference of mean cigarettes smoked per day at Baseline and Quit Date (Mean CPD at Baseline - Mean CPD at Quit Date)
Statistical Analysis 2: Comparison: Baseline (BL) vs 3-month Follow-up (3MFU); Test type: Other — A paired-samples t-test was used to evaluate smoking reduction in participants from baseline (BL) to 3-month follow-up session (3MFU); p = .067, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 11.9, 95% CI 2-sided [-1.55 to 25.35], Standard Deviation 8.45 — Mean difference represents the difference of mean cigarettes smoked per day at Baseline and 3-month follow-up. Estimated value reported is reflective of the n=4 participants that attended the 3-month follow-up session

8. Secondary Outcome: Change in Total Emotional Distress
Description: Self-reported change in emotional distress was evaluated via the 21-item, Depression, Anxiety and Stress Scale (DASS-21). The DASS-21 is composed of three self-report scales that measure the emotional states of depression, anxiety and stress. Items are rated on a Likert-type scale (0=Did not apply to me at all, to 3=Applied to me very much, or most of the time). Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items. The severity ratings are as follows Depression: Normal 0-4, Mild: 5-6, Moderate: 7-10, Severe: 11-13, Extremely Severe: 14-21. Stress: Normal: 0-7, Mild: 8-9, Moderate: 10-12, Severe: 13-16, Extremely Severe: 17-21. Anxiety: Normal: 0-3, Mild: 4-5, Moderate: 6-7, Severe: 8-9, Extremely Severe: 10-21. Total scores are computed by summing the subscales. Total scores for the DASS-21 range from 0-63. For all scales, higher scores are indicative of greater emotional distress and less change in total distress symptoms over time.
Time Frame: Week 0 (i.e., baseline), Week 5 (i.e., 2-weeks post-quit), Week 7 (i.e., 1-month post-quit) and Week 16 (i.e., 3-month follow-up)
Population: Of the N=10 participants who were eligible and attended their baseline session, n=6 attended their 2-weeks post-quit session, n=5 attended their 1-month post-quit session, n=4 attended 3-month follow-up session.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline (BL): Participants who attended their baseline session
- 2-weeks Post-quit (2W): Participants who attended their 2-weeks post-quit session
- 1-month Post-quit (1M): Participants who attended their 1-month post-quit session
Arm/Group | Baseline (BL) | 2-weeks Post-quit (2W) | 1-month Post-quit (1M) | 3-month Follow-up (3MFU)
Number analyzed (Participants) | 10 | 6 | 5 | 4
score on a scale
  DASS-21 Total score | 39.9 (14.0) | 23.5 (12.85) | 12.2 (3.11) | 13.75 (6.55)
  DASS-21 Depression score | 11.5 (4.74) | 5.0 (2.76) | 3.0 (2.23) | 4.0 (2.71)
  DASS-21 Anxiety score | 11.7 (4.39) | 5.3 (1.75) | 2.8 (1.64) | 3.5 (1.29)
  DASS-21 Stress score | 16.7 (6.03) | 13.17 (10.07) | 6.4 (2.07) | 6.25 (2.98)
Statistical Analysis 1: Comparison: Baseline (BL) vs 2-weeks Post-quit (2W); Test type: Other — A paired-samples t-test was conducted to examine the difference in the DASS-21 total score from baseline (BL) to 2-weeks post-quit (2W); p = .010, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 19.67, 95% CI 2-sided [7.17 to 32.17], Standard Deviation 11.91 — Mean difference represents the difference of mean DASS-21 total scores at Baseline and 2-weeks post-quit. Estimated value reported is reflective of the n=6 participants that attended the 2-weeks post quit session
Statistical Analysis 2: Comparison: Baseline (BL) vs 1-month Post-quit (1M); Test type: Other — A paired-samples t-test was conducted to examine the difference in DASS-21 Total scores from baseline (BL) to 1-month post-quit (1M); p = .027, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 31.2, 95% CI 2-sided [5.88 to 56.52], Standard Deviation 20.4 — Mean difference represents the difference of mean DASS-21 total scores at Baseline and 1-month post-quit. Estimated value reported is reflective of the n=5 participants that attended the 1-month post-quit session
Statistical Analysis 3: Comparison: Baseline (BL) vs 3-month Follow-up (3MFU); Test type: Other — A paired-samples t-test was conducted to evaluate the difference in DASS-21 total scores from baseline (BL) to 3-month follow up (3MFU); p = .045, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 25.75, 95% CI 2-sided [1.09 to 50.41], Standard Deviation 15.5 — Mean difference represents the difference of mean DASS-21 total scores at Baseline and 3-month follow-up. Estimated value reported is reflective of the n=4 participants that attended the 3-month follow-up session

ADVERSE EVENTS:
Time Frame: Baseline (i.e. Week 0), End of Treatment (i.e. Week 7, 1-month post-quit), 3-month follow-up (i.e. Week 16)
Arm/Group | Enrolled
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT03972137/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT03972137/Prot_SAP_003.pdf